CLINICAL TRIAL: NCT07396987
Title: Boosting Referrals to Asthma Specialists for Patients Seen at the Emergency Room for an Asthma Exacerbation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Carlos Cardet (Other)
Collaborators: Tampa General Hospital (Other); University of South Florida (Other); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Juan Carlos Cardet, Associate Professor - Research, College of Medicine Internal Medicine, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ORIGINS
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Asthma Attack; Asthma Control; Asthma Exacerbations; Asthma
Keywords: asthma; asthma exacerbation; asthma control; inhaled corticosteroid; Long-Acting Beta-Agonist; Long-Acting Muscarinic Antagonist; Emergency Room; Asthma Control Test; Medication Adherence Report Scale for Asthma; Asthma Symptom Utility Index; barriers to care; social determinants of health; access to care; telehealth; telemedicine
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will receive two components:
  1. Emergency Room (ER) staff will directly contact the asthma specialist's scheduling team to arrange a follow-up appointment within 1-3 weeks.
  2. The follow-up appointment will be conducted via telehealth (including phone calls) to assess follow-up care and asthma control of all participants.
  Both Arms:
  • All participants will be offered a prescription for twice-daily ICS/LABA (fluticasone/salmeterol) controller therapy at ER discharge after signing informed consent. These medications are standard of care for asthma.
  Asthma-related surveys and study-specific questionnaires, "medication side effects (open-ended)" and "follow-up care questions" will be administered during the ER visit and again at the 3-month follow-up phone call.
  Interventions: Behavioral: ER-Initiated Telehealth Referral
- Usual Care Arm (No Intervention): Participants will receive an EMR-based referral to an outpatient allergy clinic, with the option of a telehealth or in-person visit at their discretion. This referral will be offered during the 3-month follow-up phone call to ensure clinical equipoise.
  Both Arms:
  • All participants will be offered a prescription for twice-daily ICS/LABA (fluticasone/salmeterol) controller therapy at ER discharge after signing informed consent. These medications are standard of care for asthma.
  Asthma-related surveys and study-specific questionnaires, "medication side effects (open-ended)" and "follow-up care questions" will be administered during the ER visit and again at the 3-month follow-up phone call.

INTERVENTIONS:
Behavioral: ER-Initiated Telehealth Referral — Participants assigned to the intervention arm will receive an asthma specialist follow up appointment that is scheduled directly from the emergency department before discharge. Emergency department staff will contact the specialist clinic to arrange a telehealth visit within 1-3 weeks. The telehealth visit will address asthma symptoms, medication use, and follow-up care needs. All participants, including those in the intervention arm, will be offered a prescription for standard inhaled corticosteroid/long-acting beta-agonist controller therapy at discharge. The intervention focuses on improving access to specialist care through proactive scheduling and telehealth delivery.
  Arms: Intervention Arm

SUMMARY:
This study is testing a new way to help adults with asthma get follow up care after an emergency room (ER) visit for an asthma attack. Many people who come to the ER for asthma never see an asthma specialist afterward, even though specialists can offer treatments such as advanced inhalers or biologic medicines that may prevent future attacks.

The study will compare two approaches. One group will receive a telehealth appointment with an asthma specialist that is scheduled for them before they leave the ER. The other group will receive the usual care, which typically includes a standard referral but no scheduled appointment. All participants will be offered a prescription for standard controller medication at discharge.

The main question the study aims to answer is whether arranging a telehealth visit directly from the ER increases the number of patients who complete a follow up appointment with an asthma specialist within three months. The study will also look at whether this approach improves asthma control, reduces repeat ER visits, and helps patients better understand and use their asthma medications.

This research may help identify a practical way to improve access to asthma specialists and reduce the burden of asthma for patients who frequently rely on emergency care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Asthma diagnosis ≥1 year
* Seen in ER for asthma exacerbation
* Persistent asthma on controller therapy
* ≥1 asthma exacerbation in prior year

We will allow for current smokers, vapers and cannabis users as long as they have not been diagnosed with COPD and have a smoking history <10 pack-years.

We will allow for COPD as long as they are:

1. never smokers/vapers/cannabis users; or
2. former or current smokers/vapers/cannabis users with normal pulmonary function tests (PFT; FEV1/FVC ratio of >70%) within 12 months of enrollment and a smoking history <10 pack-years; or
3. current or former smoker/vapers/cannabis users with obstruction on PFTs (FEV1/FVC ratio of <70%) but who demonstrate BOTH >10% acute bronchodilator reversibility AND a normal diffusing capacity both within 12 months of enrollment (stricter criteria than those used in the PREPARE trial (15) and a smoking history <10 pack-years.

Exclusion Criteria:

* Patients who have seen an asthma specialist (allergist or pulmonologist) for asthma in the past 2 years
* Diagnosis of other pulmonary diseases (e.g., COPD, interstitial lung disease, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Completing an Asthma Specialist Follow-Up Visit Within 3 Months After Emergency Department Discharge | Within 3 months after emergency department discharge
  Completion of an asthma specialist follow-up visit will be assessed using documentation in the electronic health record. A visit will be counted if the record shows that the participant completed a telehealth or in-person appointment with an asthma specialist within 3 months after the emergency department discharge. The outcome will be reported as the proportion of participants in each study arm who completed a qualifying specialist visit during the 3-month follow-up period.

SECONDARY OUTCOMES:
Proportion of Participants Experiencing an Additional Asthma Exacerbation Within 3 Months After Emergency Department Discharge | Within 3 months after emergency department discharge
  A secondary asthma exacerbation will be identified using electronic health record documentation of an asthma related emergency department visit, hospitalization, or need for systemic corticosteroids within 3 months after discharge. The outcome will be reported as the proportion of participants experiencing at least one exacerbation.
Change in Asthma Control Test (ACT) Score From Baseline to 3 Months | Within 3 months after emergency department discharge
  Asthma control will be assessed using the Asthma Control Test (ACT), a validated 5 item questionnaire with scores ranging from 5 to 25, where higher scores indicate better asthma control. The outcome will be reported as the change in ACT score from baseline to 3 months.
Improvement in quality of life via Asthma Symptom Utility Index (ASUI) | Within 3 months after emergency department discharge
  Measure will be taken through the Asthma Symptom Utility Index (ASUI), an 11-item questionnaire, adminstered during the ER visit and at three month follow up. The summary score is continuous, ranging from 0 to 1.
Adherence to Controllers (MARS5) | Within 3 months after emergency department discharge
  The MARS5 questionnaire is a 5-item self-report questionnaire assessing adherence to treatments like controllers, scoring from 5 (low) to 25 (high). It measures behaviors such as forgetting, altering, stopping, or skipping doses, with a score of or often indicating high adherence.
Repeat ER visits | Within 3 months after emergency department discharge
  Repeat ER visits for asthma
Asthma hospitalizations | Within 3 months after emergency department discharge
  Participants who are hospitalized for asthma.

OTHER OUTCOMES:
Patient subjective experience with asthma care after ER visit, assessed using a structured qualitative interview | Within 3 months of emergency department discharge
  This outcome will be assessed using a semi structured qualitative interview developed for this study, conducted at the 3 month follow up call. The tool includes open ended questions designed to qualitatively evaluate participant's subjective asthma care experience after the ER visit. Themes assessed include:
  * Confusion about the asthma controller therapy regimen
  * Biologic therapy initiation or recommendations
  * Controller medication use
  * Diagnostic workup understanding
  * Whether participants report being offered information about clinical research opportunities in asthma
  Responses will be transcribed and thematically coded. The unit of measure will be the number of participants expressing each predefined theme.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Cardet, MD, Principal Investigator — University of South Florida

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: The IPD and supporting information will be available for 15 years after the conclusion of this study.
Access Criteria: Data will be labeled with unique deidentified codes. Only Tampa General Hospital and University of South Florida staff authorized on this or future related research would have access to the data. There are no specimens being collected for this study.
  Release requests will be submitted to the Principal Investigator (PI) at:
  Dr. Juan Carlos Cardet, MD For IRB Study # STUDY009146 409 Bayshore Blvd, 5th Floor Tampa, FL 33606
  Requests should include the following information:
  * Purpose of the data use
  * Description of the data requested
  * Intended future research or analysis
  * Any associated agreements (e.g., Data Use Agreements or Material Transfer Agreements)
  Approvals Required:
  • PI Approval: The PI must review and approve the release request.
  Who Can Obtain Data:
  * Qualified Researchers: Only individuals with appropriate credentials and institutional affiliations may receive data.
  * External Collaborators: Must be covered under a formal agreement (e.g., IRB reliance agreement, data

REFERENCES:
- [Background] Israel E, Cardet JC, Carroll JK, Fuhlbrigge AL, She L, Rockhold FW, Maher NE, Fagan M, Forth VE, Yawn BP, Arias Hernandez P, Kruse JM, Manning BK, Rodriguez-Louis J, Shields JB, Ericson B, Colon-Moya AD, Madison S, Coyne-Beasley T, Hammer GM, Kaplan BM, Rand CS, Robles J, Thompson O, Wechsler ME, Wisnivesky JP, McKee MD, Jariwala SP, Jerschow E, Busse PJ, Kaelber DC, Nazario S, Hernandez ML, Apter AJ, Chang KL, Pinto-Plata V, Stranges PM, Hurley LP, Trevor J, Casale TB, Chupp G, Riley IL, Shenoy K, Pasarica M, Calderon-Candelario RA, Tapp H, Baydur A, Pace WD. Reliever-Triggered Inhaled Glucocorticoid in Black and Latinx Adults with Asthma. N Engl J Med. 2022 Apr 21;386(16):1505-1518. doi: 10.1056/NEJMoa2118813. Epub 2022 Feb 26. PMID: 35213105; PMCID: PMC10367430.
- [Background] Ugalde IC, Ratigan A, Merriman C, Cui J, Ericson B, Busse P, et al. Preference for and impact of telehealth vs inperson asthma visits among Black and Latinx adults. Ann Allergy Asthma Immunol. 2023;131(5):614-27 e2.
- [Background] Maldonado-Puebla M, Akenroye A, Busby J, Cardet JC, Louisias M. Pharmacoequity in Allergy-Immunology: Disparities in Access to Medications for Allergic Diseases and Proposed Solutions in the United States and Globally. J Allergy Clin Immunol Pract. 2024;12(2):272-80.
- [Background] Patadia R, Casale TB, Fowler J, Patel S, Cardet JC. Advancements in biologic therapy in eosinophilic asthma. Expert Opin Biol Ther. 2024;24(4):251-61.
- [Background] Inselman JW, Jeffery MM, Maddux JT, Shah ND, Rank MA. Trends and Disparities in Asthma Biologic Use in the United States. J Allergy Clin Immunol Pract. 2020;8(2):549-54 e1.
- [Background] National Asthma E, Prevention P. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007;120(5 Suppl):S94-138.
- [Background] Carr T, Tkacz J, Chung Y, Ambrose CS, Spahn J, Rane P, et al. Gaps in Care Among Uncontrolled Severe Asthma Patients in the United States. J Allergy Clin Immunol Pract. 2024;12(7):1775-82 e2.
- [Background] Ortega H, Bharmal N, Khatri S. Primary care referral patterns for patients with asthma: analysis of real-world data. J Asthma. 2023;60(3):609-15.
- [Background] Yaghoubi M, Adibi A, Safari A, FitzGerald JM, Sadatsafavi M. The Projected Economic and Health Burden of Uncontrolled Asthma in the United States. Am J Respir Crit Care Med. 2019;200(9):1102-12.
- [Background] Nurmagambetov T, Kuwahara R, Garbe P. The Economic Burden of Asthma in the United States, 2008-2013. Ann Am Thorac Soc. 2018;15(3):348-56.
- [Background] Dean BB, Calimlim BC, Sacco P, Aguilar D, Maykut R, Tinkelman D. Uncontrolled asthma: assessing quality of life and productivity of children and their caregivers using a cross-sectional Internet-based survey. Health Qual Life Outcomes. 2010;8:96.
- [Background] Most Recent National Asthma Data: Centers for Disease Control and Prevention; 2022 [Available from: https://www.cdc.gov/asthma/most_recent_national_asthma_data.htm.
- [Background] Taunk ST, Cardet JC, Ledford DK. Clinical implications of asthma endotypes and phenotypes. Allergy Asthma Proc. 2022;43(5):375-82.
- [Background] Ishmael L, Casale T, Cardet JC. Molecular Pathways and Potential Therapeutic Targets of Refractory Asthma. Biology (Basel). 2024;13(8).
- [Background] Buhl R, Bel E, Bourdin A, Davila I, Douglass JA, FitzGerald JM, et al. Effective Management of Severe Asthma with Biologic Medications in Adult Patients: A Literature Review and International Expert Opinion. J Allergy Clin Immunol Pract. 2022;10(2):422-32.